CLINICAL TRIAL: NCT06325254
Title: A Multicenter, Retrospective Clinical Study on the Clinical Characteristics of Metabolic Associated Fatty Liver Disease
Brief Title: Clinical Characteristics of Metabolic Associated Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jie Li, Principal investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: MAFLD
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Metabolic Associated Fatty Liver Disease; Clinical Features
Keywords: Metabolic associated fatty liver disease; Clinical features

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic associated fatty liver disease (MAFLD), which can lead to liver fibrosis, cirrhosis, liver failure and even hepatocellular carcinoma, poses a significant burden on society. With the improvement of living standards and changes in dietary habits, MAFLD patients show a younger and increasing trend, but there is still no specific drug. The clinical features and prognosis of MAFLD may be different with different metabolic disorder phenotypes and treatment measures. Therefore, further systematic study of the clinical characteristics and prognosis of MAFLD patients will be of great significance for the formulation of corresponding clinical prevention and treatment strategies.

DETAILED DESCRIPTION:
Metabolic associated fatty liver disease (MAFLD), which can lead to liver fibrosis, cirrhosis, liver failure and even hepatocellular carcinoma, poses a significant burden on society. With the improvement of living standards and changes in dietary habits, MAFLD patients show a younger and increasing trend, but there is still no specific drug. The clinical features and prognosis of MAFLD may be different with different metabolic disorder phenotypes and treatment measures. Therefore, further systematic study of the clinical characteristics and prognosis of MAFLD patients will be of great significance for the formulation of corresponding clinical prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older;
2. MAFLD patients

Exclusion Criteria:

1. malignant tumors;
2. mental illness, severe impairment of cardiopulmonary function, severe renal insufficiency, severe infections, and cerebrovascular accidents;
3. received liver or other organ transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MAFLD patients
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics and follow-up outcomes of MAFLD patients | 480 weeks
  1. Clinical characteristic related indicators: height (m), weight (kg), waist circumference (cm), previous history (T2DM, HT, dyslipidemia), SBP (mmHg), DBP (mmHg), alcohol intake (g/week), smoking, blood routine [WBC (109/L), Hb (g/L), PLT (109/L)], CRP (mg/L), biochemical indicators [TB (umol/L), ALB (g/L), ALT (U/L), AST (U/L), ALP (U/L), GGT (U/L), TC (mmol/L), TG (mmol/L), HDL (mmol/L), LDL (mmol/L)], blood glucose indicators [FBG (mmol/L), PBG (mmol/L), HA1c (%)], coagulation [PT (s), INR], AFP (ng/ml), transient elastography [LSM (Kpa), ACP (dB/m)], liver CT/MRI/B type ultrasound.
  2. Follow up outcome data: mortality and causes of death, incidence of complications (ascites, variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, intrahepatic and extrahepatic malignancies, infection, cardiovascular and cerebrovascular diseases, or all-cause mortality).

SECONDARY OUTCOMES:
Clinical characteristics and follow-up outcomes of MAFLD patients under different subgroups | 480 weeks
  1. Subgroups: Age (<40 years and ≥40 years), gender (male and female), steatosis stage according to CT/MRI/B type ultrasound (Mild, moderate, and severe), and MASH status (non-MASH and MASH)
  2. Clinical characteristic related indicators: height (m), weight (kg), waist circumference (cm), previous history (T2DM, HT, dyslipidemia), SBP (mmHg), DBP (mmHg), alcohol intake (g/week), smoking, WBC (109/L), Hb (g/L), PLT (109/L), TB (umol/L), ALB (g/L), ALT (U/L), AST (U/L), ALP (U/L), GGT (U/L), TC (mmol/L), TG (mmol/L), HDL (mmol/L), LDL (mmol/L), FBG (mmol/L), PBG (mmol/L), HA1c (%), PT (s), INR, AFP (ng/ml), transient elastography [LSM (Kpa), ACP (dB/m)], liver CT/MRI/B type ultrasound, liver histology.
  3. Follow up outcome data: mortality and causes of death, incidence of complications.
Baseline clinical characteristics MAFLD patients | 0 weeks
  Clinical characteristic related indicators: height (m), weight (kg), waist circumference (cm), previous history (T2DM, HT, dyslipidemia), SBP (mmHg), DBP (mmHg), alcohol intake (g/week), smoking, blood routine [WBC (109/L), Hb (g/L), PLT (109/L)], CRP (mg/L), biochemical indicators [TB (umol/L), ALB (g/L), ALT (U/L), AST (U/L), ALP (U/L), GGT (U/L), TC (mmol/L), TG (mmol/L), HDL (mmol/L), LDL (mmol/L)], blood glucose indicators [FBG (mmol/L), PBG (mmol/L), HA1c (%)], coagulation [PT (s), INR], AFP (ng/ml), transient elastography [LSM (Kpa), ACP (dB/m)], liver CT/MRI/B type ultrasound.
Risk factors for progression to cirrhosis and hepatocellular carcinoma | 480 weeks
  Risk factors for progression to cirrhosis and hepatocellular carcinoma in MAFLD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China